CLINICAL TRIAL: NCT00194493
Title: Computerized Assessment for Patients With Cancer
Acronym: ESRA-C
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, Donna Berry, PhD, RN, FAAN, ACON, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APP00000089; R01NR008726 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Neoplasms
Keywords: Cancer; Quality of Life; Signs and Symptoms; Computers; Patient-Reported Outcomes
MeSH Terms: conditions — Neoplasms; Signs and Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Patient's clinician receives graphical report of patient-reported symptoms and quality of life issues.
  Interventions: Behavioral: ESRA-C
- 2 (No Intervention)

INTERVENTIONS:
Behavioral: ESRA-C — Graphical summary of patient symptoms and quality of life
  Arms: 1

SUMMARY:
The traditional procedure for cancer symptom and quality of life instrument administration is a paper questionnaire completed by the patient or research participant. The use of standardized, patient report instruments as routine assessment in clinical cancer care has been promoted, but infrequently reported and the utilization rate is low. Barriers to clinical use include the personnel cost of data collection, management of written questionnaires and the clinicians' unfamiliarity with the nature of the queries and numerical scale scores. Web-based electronic technology now has been developed and tested for feasibility using touchscreen, notebook computers and the computerized assessment program, a screening assessment providing usable and easily interpreted graphic output to cancer clinicians. The purpose of this study is to design and evaluate the clinical integration of the web-based computerized assessment in a major, multi-disciplinary academic medical center and cancer center. Consecutive outpatients who are evaluated for cancer therapy in each of the 2 setting sites, the University of Washington Medical Center and the Seattle Cancer Care Alliance, are able to communicate in English (or through one of the many interpreters available at the institutions), and are competent to understand the study information and give informed consent will be invited to participate. Clinicians caring for the patients in the sample will be invited to participate in evaluating the organizational impact. We will compare the outcomes of conducting assessment in the usual practices and procedures to the outcomes of using the computerized assessment program: appropriateness of referrals, efficiency, and usability. The computerized assessment will be completed prior to each participant's visit with the clinician, conducted at the first clinic visit, during the 4-6th week of treatment and again at a 30 day follow up visit. Graphical output will be immediately available to clinicians. Descriptive, comparative statistics will be used to evaluate the impact of the screening and longitudinal assessments.

DETAILED DESCRIPTION:
Patients with cancer, across a wide range of diagnoses and stages, have a high incidence of symptoms that may greatly impact quality of life. The consequences of inadequate symptom assessment and management are profound, complex, and can be overwhelming to patients and their caregivers. However, clinicians are faced too often with shrinking resources, removing opportunities for comprehensive, interpersonal interactions with patients. The patient's experience, particularly symptoms and quality of life (QOL) concerns, reported in a reliable and systematic way, is an essential component of the information on which a complete clinical assessment, diagnosis and treatment plan is based. Computer technology has been developed for patient self-reporting of symptom and QOL data using validated survey instruments delivered on notebook computers, personal digital assistants, and over the Web. Not only do these devices eliminate the usual steps of abstracting patient interview data and/or keying in marked responses, but the interfaces also permit customized, confidential and private assistance with answering queries more completely. While the reports are few, the results are positive: data integrity is enhanced by the computerized assessment, and patients prefer, and are easily able to complete the computerized versions. Furthermore, computerized screening procedures have demonstrably enhanced communication between clinicians and patients and successfully identified psychologically distressed patients with cancer.

* Clinicians and researchers developed and pilot-tested the ESRA-C prototype in 2000/2001 at the University of Washington Medical Center Cancer Center. The successful implementation was published in 2004 in the Oncology Nursing Forum. [8]
* The purpose of this new randomized trial is to evaluate the clinical use of our web-based ESRA-C throughout the Seattle Cancer Care Alliance.
* Two patients per month per team (Transplant) or per provider (Radiation Oncology, Medical Oncology) will be enrolled in this study.
* Patients will use the system to self-assess their symptoms and QOL at 2 time points, before (T1) and after treatment (T2)
* At the second, on-treatment assessment, the intervention group patients will have a color-graphic summary of their answers from both T1 and T2 delivered to the clinical team before the clinic visit with the patient.
* Both intervention and control participants will have the T2 clinic visit audio-recorded. Clinician data will be anonymously entered and audio-files destroyed.
* Using chart reviews we will abstract any notations, therapies ordered, prescriptions written and referrals made, relevant to symptoms and quality of life issues. This will be documented without clinician identifiers.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Cancer

Exclusion Criteria:

* Less than 18 years of age
* Non-english speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1058 (Actual)
Dates: Start 2005-04; Primary Completion 2007-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Frequency of QOL and symptom topics being addressed in audiotaped patient/clinician visits | Study end
Frequency of QOL and symptom information being documented by clinician in the medical record within 24 hours | Study end
Frequency of appropriate symptom interventions recommended by clinicians and documented in the medical record | Study end
Frequency of appropriate referrals to specialty or support services subsequent to assessment. | Study end

SECONDARY OUTCOMES:
Process Variables (Efficiency process,Usability process) | Study end
Clinical Significance (Score change over time,Magnitude of change, Response shift) | Study end

CONTACTS AND LOCATIONS:
Overall Officials: Donna L Berry, PHD RN, Principal Investigator — School of Nursing, University of Washington
Locations (2):
- United States (2):
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington